CLINICAL TRIAL: NCT06752980
Title: The Effect of Eye Mask and Earplugs on Sleep Quality and Delirium in Coronary Artery Bypass Graft Patients: A Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeliha Birer, Nurse, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NecmettinEU-SBF-ZB-01
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Surgical Procedures
Keywords: Cardiovascular surgical procedures, Delirium, Sleep
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eye Mask and Earplugs (Experimental): On the 1st, 2nd and 3rd postoperative day, the experimental group will be given the intervention reserved during their night sleep, using eye patches and earplugs.
  On the 2nd, 3rd and 4th postoperative day, repeated monitoring will be performed using RCUÖ and Nu-DESC.
  Patients who wish to leave the study at any stage, do not receive the reserved intervention or die during the monitoring will be excluded from the study.
- Earplugs (Experimental): The reserved intervention will be applied during the night sleep with earplugs on the 1st, 2nd and 3rd day group after the surgery.
  Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th days after the surgery.
  Patients who want to leave at any stage of the study, do not receive the reserved intervention or die during the monitoring will be excluded from the study.
- Eye Mask (Experimental): The intervention allocated during night sleeps with Eye Mask applied on the 1st, 2nd and 3rd days after the surgery will be applied.
  Repeated monitoring will be done using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th days after the surgery.
  Patients who want to leave at any stage of the study, do not perform the allocated intervention or die during the follow-up will be excluded from the study.
  Interventions: Other: Eye mask
- no mask no earblugs (No Intervention): No intervention will be performed on the 1st, 2nd and 3rd postoperative day.
  Repeated monitoring will be performed on the 2nd, 3rd and 4th postoperative day using RCUÖ and Nu-DESC.
  Patients who wish to leave the study at any stage, who do not perform the intervention, or who die during follow-up will be excluded from the study.

INTERVENTIONS:
Other: Eye mask — The three experimental groups (eye patch group, earplug group, eye patch and earplug group applied together) will be given a separate intervention during their night sleep on the 1st, 2nd and 3rd postoperative day. Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th postoperative days.
  Arms: Eye Mask
Other: Earplugs — The three experimental groups (eye patch group, earplug group, eye patch and earplug group applied together) will be given a separate intervention during their night sleep on the 1st, 2nd and 3rd postoperative day. Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th postoperative days.
Other: Eye Mask and Earplugs — The three experimental groups (eye patch group, earplug group, eye patch and earplug group applied together) will be given a separate intervention during their night sleep on the 1st, 2nd and 3rd postoperative day. Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th postoperative days.

SUMMARY:
Coronary artery bypass grafting is the most commonly performed surgical procedure among cardiovascular diseases. Nursing care for patients undergoing cardiac surgery involves a process that includes preoperative preparation and subsequent close monitoring of neurological, cardiac, respiratory, vascular status, kidney function, and pain. Sleep disturbances are observed after cardiac surgery. Sleep plays a critical role in the body's maintenance, repair, and renewal processes. Improved sleep can reduce patient agitation and decrease the risk of delirium. The presence of delirium leads to increased care requirements and prolonged hospital stays, which in turn raises hospital costs. Enhancing sleep quality and preventing delirium after surgery have positive effects on clinical patient outcomes. This study is designed to determine the effects of using eye masks and/or earplugs on sleep quality and delirium in patients undergoing coronary artery bypass grafting during nighttime sleep. This research is a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

-Patients who voluntarily agree to participate in the study

* Those who have undergone coronary artery bypass graft surgery
* Those between the ages of 18-79
* Those who are cooperative and oriented
* Those who are literate
* Those who speak Turkish
* Those whose initial delirium scale score (Nu-DECS) is less than 2
* Those whose Glasgow coma scale score is >13 will be included in the study.

Exclusion Criteria:

* • Patients diagnosed with sleep disorders,

  * Those using sleeping pills,
  * Those who have a habit of using an eye patch while sleeping,
  * Those who were not transferred to the clinic on the first day after surgery and whose treatment continues in the intensive care unit,
  * Those who develop complications and/or need to be re-operated,
  * Those who need treatment other than routine treatment,
  * Patients with hearing or vision problems will be excluded.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Scale | Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th days after surgery.
  The RCUS was developed by Richards and colleagues (1987) to assess sleep. The RCUS includes six items (sleep depth, time to fall asleep, frequency of awakenings, time to remain awake when awakened, quality of sleep, and ambient noise level). Each item is rated using a 0-100 visual analog scale. The total score is obtained by dividing the individual items by their numbers: 0 represents the worst sleep, 100 the best sleep. As the score obtained from the scale increases, the sleep quality of the patients also increases. The RCUS provides a short, applicable, comprehensive, and simple tool for assessing sleep quality in the intensive care unit and is the most common. The Cronbach α value of the scale was found to be 0.82. The validity and reliability study of the scale in our country was conducted by Karaman Özlü and Özer (2015). The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.91.
Nursing Delirium Screening Scale- Nu-DESC | Repeated monitoring will be performed using RCUÖ and Nu-DESC on the 2nd, 3rd and 4th days after surgery.
  The scale consists of five items. These are; disorientation, inappropriate behavior, inappropriate communication, illusion-hallucination and slowness in psychomotor behavior. It is critical that all subtypes can be detected in an effective delirium diagnosis. Among the items in Nu-DESC, it is thought that hypoactive delirium is detected more successfully with the item that evaluates psychomotor slowness. Each item in the scale takes a value between 0 and 2 points and the total score varies between 0 and 10. Two points and above indicate delirium. The evaluation time is approximately one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Saide Faydalı, Study Director — Necmeetin Erbakan University
Locations (1):
- Necmettin Erbakan Universıty, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilic G, Kav S. Effect of using eye masks and earplugs in preventing delirium in intensive care patients: A single-blinded, randomized, controlled trial. Nurs Crit Care. 2023 Sep;28(5):698-708. doi: 10.1111/nicc.12901. Epub 2023 May 3. PMID 37138379